CLINICAL TRIAL: NCT03841331
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy, Safety, and Tolerability of Serlopitant for the Treatment of Chronic Pruritus of Unknown Origin
Brief Title: Study of the Efficacy, Safety, and Tolerability of Serlopitant for the Treatment of Chronic Pruritus of Unknown Origin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTI-117
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Results first posted 2020-09-23 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Pruritus
Keywords: Pruritus
MeSH Terms: conditions — Pruritus | interventions — serlopitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 5 mg Serlopitant Tablets (Experimental): Serlopitant Tablets
  Interventions: Drug: 5 mg Serlopitant Tablets
- 5 mg Placebo Tablets (Placebo Comparator): Placebo Tablets
  Interventions: Drug: Matching Placebo Tablets

INTERVENTIONS:
Drug: 5 mg Serlopitant Tablets — Serlopitant Tablets
  Other Names: VPD-737
  Arms: 5 mg Serlopitant Tablets
Drug: Matching Placebo Tablets — Placebo Tablets
  Arms: 5 mg Placebo Tablets

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy, Safety, and Tolerability of Serlopitant for the Treatment of Chronic Pruritus of Unknown Origin

ELIGIBILITY:
Inclusion:

* Male or female, age 18 years or older at consent.
* The subject must have ongoing chronic pruritus
* The subject's pruritus is assessed by the investigator to be of unknown origin at baseline.
* Worst-Itch Numeric Rating Scale (WI-NRS) score in the 24-hour period prior to the Screening visit, and average weekly WI-NRS score in each of the 2 weeks prior to Baseline visit indicating an appropriate pruritus level for the study.
* The pruritus must have been unresponsive to prior treatment with emollients.
* The subject's pruritus must be present on multiple segments of the body
* Willing and able to complete daily eDiary entries within a consistent timeframe for the duration of the study
* All females who are of childbearing potential must be willing to practice highly effective contraception and not be pregnant or nursing
* Willing to comply with study visits and study related requirements including providing written informed consent.
* Adequate cognitive and physical ability, in the investigator's opinion, to comply with study visits and study related requirements including providing written informed consent

Exclusion

* Prior treatment with any NK1-receptor antagonists
* Known dermatologic or systemic condition(s), other than dry skin, that is considered by the investigator to be the primary cause of current pruritus.
* Untreated or inadequately treated thyroid, adrenal, or pituitary disease or nodules, or history of thyroid malignancy.
* Use of an excluded therapy within 3 weeks prior to randomization
* Treatment with any investigational therapy within 3 weeks prior to randomization.
* Serum creatinine, total bilirubin, alanine aminotransferase or aspartate aminotransferase > 2.5 times the upper limit of normal during screening.
* History of malignancy within 3 years prior to randomization, with the (actinic keratosis, non-metastatic cutaneous squamous cell carcinoma, basal cell carcinoma of skin).
* Any known major psychiatric diagnosis that would impact the subject's ability to complete the study
* Suicidal ideation within 3 years prior to randomization, or any history of suicide attempt.
* Known use of recreational drugs.
* Documented history of parasitic infection, including skin parasites such as scabies, within 12 weeks prior to randomization.
* Presence of clinically significant dementia, intellectual impairment, or any medical condition or disability that, in the investigator's opinion, could interfere with the assessment of safety or efficacy in this trial or compromise the safety of the subject.
* History of hypersensitivity to serlopitant or any of its components.
* Planned or anticipated major surgical procedure or other activity that would interfere with the subject's ability to comply with protocol-mandated assessments (e.g. extended international travel) during the subject's participation in the study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-01-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - Study Site 221, Hot Springs, Arkansas
  - Study Site 823, Bakersfield, California
  - Study Site 204, Fremont, California
  - Study Site 803, Los Angeles, California
  - Study Site 820, Centennial, Colorado
  - Study Site 804, Denver, Colorado
  - Study Site 811, Aventura, Florida
  - Study Site 801, Jacksonville, Florida
  - Study Site 807, Miami, Florida
  - Study Site 331, Miami, Florida
  - Study Site 824, Sarasota, Florida
  - Study Site 818, West Palm Beach, Florida
  - Study Site 349, Savannah, Georgia
  - Study Site 814, Indianapolis, Indiana
  - Study Site 808, Brighton, Massachusetts
  - Study Site 822, Rolla, Missouri
  - Study Site 371, Saint Joseph, Missouri
  - Study Site 817, St Louis, Missouri
  - Study Site 821, Bellevue, Nebraska
  - Study Site 813, Las Vegas, Nevada
  - Study Site 387, Las Vegas, Nevada
  - Study Site 816, Morristown, New Jersey
  - Study Site 121, Ocean Township, New Jersey
  - Study Site 507, Brooklyn, New York
  - Study Site 802, The Bronx, New York
  - Study Site 341, High Point, North Carolina
  - Study Site 810, Raleigh, North Carolina
  - Study Site 524, Dublin, Ohio
  - Study Site 116, Portland, Oregon
  - Study Site 522, Pittsburgh, Pennsylvania
  - Study Site 345, Johnston, Rhode Island
  - Study Site 815, Warwick, Rhode Island
  - Study Site 805, Nashville, Tennessee
  - Study Site 365, Austin, Texas
  - Study Site 120, Dallas, Texas
  - Study Site 819, Fort Worth, Texas
  - Study Site 359, Pflugerville, Texas
  - Study Site 809, San Antonio, Texas
  - Study Site 217, Norfolk, Virginia
  - Study Site 806, Spokane, Washington
  - Study Site 812, Walla Walla, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 41 sites in US from 22 January 2019 to 21 January 2020. All subjects who met the study entry criteria were randomized in a 1:1 ratio to receive daily oral doses of serlopitant 5 mg or placebo.
Pre-assignment Details: During the screening period (3 weeks), all subjects were evaluated for eligibility and assessed for conditions associated with chronic pruritus. Subjects were to complete an electronic diary (eDiary) at the Screening visit.
Groups:
- Placebo: Randomized subjects received daily oral doses of placebo following an initial 3-tablet loading dose on Day 1. Starting on Day 2, subjects took 1 tablet per day until the completion of the 10-week treatment period.
- Serlopitant 5 mg: Randomized subjects received daily oral doses of serlopitant 5 mg following an initial 3-tablet loading dose on Day 1. Starting on Day 2, subjects took 1 tablet per day until the completion of the 10-week treatment period.
Period: Overall Study
Arm/Group | Placebo | Serlopitant 5 mg
Started | 117 | 116
Completed | 108 | 106
Not Completed | 9 | 10
Not completed — Withdrawal by Subject | 4 | 9
Not completed — Lost to Follow-up | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Serlopitant 5 mg | Total
Number analyzed (Participants) | 117 | 116 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (12.05) | 60.7 (13.60) | 59.4 (12.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 83 | 176
  Male | 24 | 33 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 7 | 22
  White | 95 | 102 | 197
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Worst Itch Numeric Rating Scale 4-point Responder Rate at Week 10
Description: During the study, Worst Itch Numeric Rating Scale (WI-NRS) assessments was reported by the subject via eDiary. The daily NRS results were summarized. The daily results were averaged to create weekly measures.
  The Itch NRS is a validated, self-reported, instrument for measurement of itch intensity. It used a 24-hour recall period and asked subjects to rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable), higher scores indicated greater itch intensity. A subject was a 4-point responder if their change from baseline is ≤ -4 (i.e. a decrease of at least 4).
Time Frame: At Week 10
Population: Full Analysis Population: subset of subjects in the randomized population who were dispensed study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 117 | 116
Participants | 46 | 44
Statistical Analysis 1: Comparison: Placebo vs Serlopitant 5 mg; At Week 10; Test type: Superiority; p = 0.5861, Cochran-Mantel-Haenszel; Treatment Effect = -1.4, 95% CI 2-sided [-13.9 to 11.1] — 95% Wald confidence intervals for the treatment difference was used

2. Primary Outcome: WI-NRS 4-point Responder Rate at Weeks 2 4, 6, and 8
Description: as for outcome 1
Time Frame: At Weeks 2, 4, 6, and 8
Population: Full Analysis Population: subset of subjects in the randomized population who were dispensed study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 117 | 116
Participants
  Responders at Week 2 | 19 | 18
  Responders at Week 4 | 29 | 24
  Responders at Week 6 | 35 | 38
  Responders at Week 8 | 40 | 37
Statistical Analysis 1: Comparison: Placebo vs Serlopitant 5 mg; At Week 2; Test type: Superiority; p = 0.5651, Cochran-Mantel-Haenszel; Treatment Effect = -0.7, 95% CI 2-sided [-10.1 to 8.7] — 95% Wald confidence intervals for the treatment difference was used
Statistical Analysis 2: Comparison: Placebo vs Serlopitant 5 mg; At Week 4; Test type: Superiority; p = 0.7769, Cochran-Mantel-Haenszel; Treatment Effect = -4.1, 95% CI 2-sided [-14.8 to 6.7]; 95% Wald confidence intervals for the treatment difference was used
Statistical Analysis 3: Comparison: Placebo vs Serlopitant 5 mg; At Week 6; Test type: Superiority; p = 0.3285, Cochran-Mantel-Haenszel; Treatment Effect = 2.8, 95% CI 2-sided [-9.1 to 14.8] — 95% Wald confidence intervals for the treatment difference was used
Statistical Analysis 4: Comparison: Placebo vs Serlopitant 5 mg; At Week 8; Test type: Superiority; p = 0.6525, Cochran-Mantel-Haenszel; Treatment Effect = -2.3, 95% CI 2-sided [-14.4 to 9.8] — 95% Wald confidence intervals for the treatment difference was used

3. Primary Outcome: WI-NRS 3-point Responder Rate at Weeks 2, 4, 6, 8, and 10
Description: During the study, Worst Itch Numeric Rating Scale (WI-NRS) assessments was reported by the subject via eDiary. The daily NRS results were summarized. The daily results were averaged to create weekly measures.
  The Itch NRS is a validated, self-reported, instrument for measurement of itch intensity. It used a 24-hour recall period and asked subjects to rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable), higher scores indicated greater itch intensity. A subject was a 3-point responder if their change from baseline is ≤ -3 (i.e. a decrease of at least 3). Results presented below is of subjects who were a 3-point responder but not a 4-point responder.
Time Frame: At Weeks 2, 4, 6, 8, and 10
Population: Full Analysis Population: subset of subjects in the randomized population who were dispensed study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 117 | 116
Participants
  Responders at Week 2 | 6 | 6
  Responders at Week 4 | 8 | 14
  Responders at Week 6 | 15 | 10
  Responders at Week 8 | 14 | 15
  Responders at Week 10 | 13 | 16
Statistical Analysis 1: Comparison: Placebo vs Serlopitant 5 mg; At Week 2; Test type: Superiority; p = 0.4952, Cochran-Mantel-Haenszel; Treatment effect = 0.0, 95% CI 2-sided [-5.6 to 5.7] — 95% Wald confidence intervals for the treatment difference was used
Statistical Analysis 2: Comparison: Placebo vs Serlopitant 5 mg; At Week 4; Test type: Superiority; p = 0.0891, Cochran-Mantel-Haenszel; Treatment effect = 5.2, 95% CI 2-sided [-2.3 to 12.7] — 95% Wald confidence intervals for the treatment difference was used
Statistical Analysis 3: Comparison: Placebo vs Serlopitant 5 mg; At Week 6; Test type: Superiority; p = 0.8447, Cochran-Mantel-Haenszel; Treatment effect = -4.2, 95% CI 2-sided [-12.1 to 3.7] — 95% Wald confidence intervals for the treatment difference was used
Statistical Analysis 4: Comparison: Placebo vs Serlopitant 5 mg; At Week 8; Test type: Superiority; p = 0.4174, Cochran-Mantel-Haenszel; Treatment effect = 1.0, 95% CI 2-sided [-7.5 to 9.4] — 95% Wald confidence intervals for the treatment difference was used
Statistical Analysis 5: Comparison: Placebo vs Serlopitant 5 mg; At Week 10; Test type: Superiority; p = 0.2756, Cochran-Mantel-Haenszel; Treatment effect = 2.7, 95% CI 2-sided [-5.8 to 11.2] — 95% Wald confidence intervals for the treatment difference was used

4. Primary Outcome: Change From Baseline in WI-NRS at Weeks 2, 4, 6, 8, and 10
Description: During the study, Worst Itch Numeric Rating Scale (WI-NRS) assessments was reported by the subject via eDiary. The daily NRS results were summarized. The daily results were averaged to create weekly measures.
  The Itch NRS is a validated, self-reported, instrument for measurement of itch intensity. It used a 24-hour recall period and asked subjects to rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable), higher scores indicated greater itch intensity.
Time Frame: At Weeks 2, 4, 6, 8, and 10
Population: Full Analysis Population: subset of subjects in the randomized population who were dispensed study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 117 | 116
score on a scale
  Baseline (Observed value) | 8.37 (0.929) | 8.44 (0.855)
  Change from Baseline at Week 2 | -1.65 (2.115) | -1.61 (1.961)
  Change from Baseline at Week 4 | -2.41 (2.382) | -2.46 (2.349)
  Change from Baseline at Week 6 | -2.83 (2.624) | -2.94 (2.495)
  Change from Basline at Week 8 | -2.99 (2.647) | -2.97 (2.562)
  Change from Baseline at Week 10 | -3.34 (2.787) | -3.25 (2.545)
Statistical Analysis 1: Comparison: Placebo vs Serlopitant 5 mg; At Week 2; Test type: Superiority; p = 0.4409, ANOVA; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.49 to 0.57]
Statistical Analysis 2: Comparison: Placebo vs Serlopitant 5 mg; At Week 4; Test type: Superiority; p = 0.5496, ANOVA — At week 4; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.65 to 0.57]
Statistical Analysis 3: Comparison: Placebo vs Serlopitant 5 mg; At Week 6; Test type: Superiority; p = 0.6311, ANOVA; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.78 to 0.55]
Statistical Analysis 4: Comparison: Placebo vs Serlopitant 5 mg; At Week 8; Test type: Superiority; p = 0.02, ANOVA; Mean Difference (Final Values) = 0.4738, 95% CI 2-sided [-0.65 to 0.69]
Statistical Analysis 5: Comparison: Placebo vs Serlopitant 5 mg; At Week 10; Test type: Superiority; p = 0.3948, ANOVA; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.60 to 0.78]

5. Primary Outcome: Change From Baseline in Daily WI-NRS Scores Through Week 2
Description: as for outcome 4
Time Frame: Through 2 weeks
Population: Full Analysis Population: subset of subjects in the randomized population who were dispensed study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 117 | 116
score on a scale
  Baseline (observed value) | 8.37 (0.929) | 8.44 (0.855)
  Change from Baseline at Day 1 | -0.22 (0.879) | -0.09 (0.819)
  Change from Baseline at Day 2 | -0.85 (1.836) | -0.69 (1.264)
  Change from Baseline at Day 3 | -0.94 (1.788) | -0.77 (1.348)
  Change from Baseline at Day 4 | -1.16 (1.977) | -0.96 (1.459)
  Change from Baseline at Day 5 | -1.34 (2.103) | -0.99 (1.495)
  Change from Baseline at Day 6 | -1.33 (2.174) | -1.15 (1.892)
  Change from Baseline at Day 7 | -1.44 (2.331) | -1.35 (1.758)
  Change from Baseline at Day 8 | -1.35 (2.171) | -1.35 (1.746)
  Change from Baseline at Day 9 | -1.53 (2.210) | -1.35 (1.996)
  Change from Baseline at Day 10 | -1.63 (2.460) | -1.41 (2.023)
  Change from Baseline at Day 11 | -1.73 (2.333) | -1.69 (2.211)
  Change from Baseline at Day 12 | -1.67 (2.280) | -1.58 (2.247)
  Change from Baseline at Day 13 | -1.82 (2.335) | -1.75 (2.291)
  Change from Baseline at Day 14 | -1.92 (2.518) | -1.74 (2.266)

6. Primary Outcome: Change From Baseline in Worst-Itch Visual Analog Scale at Weeks 2, 4, 6, and 10
Description: The Itch Visual Analog Scale (VAS) is a validated, self-reported instrument for measurement of itch intensity. It used a 24-hour recall period and asked subjects to rate the worst intensity of their itch on a 100-mm horizontal line ranging from 0 mm (no itch) to 100 mm (worst itch imaginable). Higher scores indicated greater itch intensity. The VAS measurement were summarized in centimeters. WI-VAS assessments were reported by the subject via a paper form administered at study visits.
Time Frame: At Weeks 2, 4, 6, and 10
Population: Full Analysis Population: subset of subjects in the randomized population who were dispensed study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 117 | 116
score on a scale
  Baseline (Observed Value) | 82.09 (10.741) | 83.53 (11.941)
  Change from Baseline at Week 2 | -22.96 (27.425) | -20.52 (28.825)
  Change from Baseline at Week 4 | -27.01 (28.906) | -28.28 (29.731)
  Change from Baseline at Week 6 | -32.83 (31.046) | -30.92 (31.487)
  Change from Baseline at Week 10 | -37.64 (31.613) | -37.42 (32.986)
Statistical Analysis 1: Comparison: Placebo vs Serlopitant 5 mg; At Week 2; Test type: Superiority; p = 0.2440, ANOVA; Mean Difference (Final Values) = 2.44, 95% CI 2-sided [-4.98 to 9.87]
Statistical Analysis 2: Comparison: Placebo vs Serlopitant 5 mg; At Week 4; Test type: Superiority; p = 0.6349, ANOVA; Mean Difference (Final Values) = -1.27, 95% CI 2-sided [-9.20 to 6.65]
Statistical Analysis 3: Comparison: Placebo vs Serlopitant 5 mg; At Week 6; Test type: Superiority; p = 1.91, ANOVA; Mean Difference (Final Values) = 0.3407, 95% CI 2-sided [-6.40 to 10.23]
Statistical Analysis 4: Comparison: Placebo vs Serlopitant 5 mg; At Week 10; Test type: Superiority; p = 0.4960, ANOVA; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-8.52 to 8.97]

7. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Adverse events (AEs) were recorded to assess the safety and tolerability of repeated oral doses of serlopitant in adult subjects with chronic pruritus of unknown origin. Adverse events (AEs) and SAEs were recorded from the first study drug administration through the follow-up visit. After informed consent was signed, but prior to initiation of study drug, only SAEs considered by the investigator to be caused by a protocol-mandated intervention were collected.
Time Frame: From screening until the Follow-up (F/U) visit which occurred 35 days (+ 7 days) after the Week 10 visit or the last dose of study drug for subjects who discontinued study drug early.
Population: Safety Population - Subset of subjects who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 117 | 116
Participants
  TEAEs | 38 | 49
  TEAEs Leading to Treatment Discontinuation | 2 | 2
  TEAEs Likely Related to Study Drug | 3 | 12
  Serious TEAEs | 0 | 2

8. Secondary Outcome: Plasma Concentrations of Serlopitant and Metabolites
Description: The plasma concentrations of serlopitant and metabolites were combined with the data from other serlopitant clinical studies for population pharmacokinetic analysis.
Time Frame: At Week 10
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo | Serlopitant 5 mg
Number analyzed (Participants) | 117 | 116
nmol/L
  Met-Serl-M1/M1a | 0.2 (2.02) | 150.8 (120.33)
  Met-Serl-M2/M2a | 0.1 (0.81) | 41.6 (26.69)
  Met-Serl-M3 | 0.0 (0.46) | 60.9 (39.43)
  Serlopitant | 0.3 (3.09) | 634.6 (441.07)

ADVERSE EVENTS:
Time Frame: From screening until the Follow-up (F/U) visit which occurred 35 days (+ 7 days) after the Week 10 visit or the last dose of study drug for subjects who discontinued study drug early.
Description: Adverse events (AEs) and serious adverse events (SAEs) were recorded from the first study drug administration through the follow-up visit. After informed consent was signed, but prior to initiation of study drug, only SAEs considered by the investigator to be caused by a protocol-mandated intervention were collected.
Arm/Group | Placebo | Serlopitant 5 mg
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/116
Serious Adverse Events (participants affected / at risk) | 0/117 | 2/116
Other Adverse Events (participants affected / at risk) | 1/117 | 12/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=117) | Serlopitant 5 mg (N=116)
Intracranial mass (Nervous system disorders) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=117) | Serlopitant 5 mg (N=116)
Diarrhoea (Gastrointestinal disorders) | 0 | 8
Somnolence (Nervous system disorders) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT03841331/Prot_002.pdf
  • Statistical Analysis Plan (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT03841331/SAP_003.pdf